CLINICAL TRIAL: NCT06784713
Title: DIFFERENT SARS-COV-2 VARIANTS' EFFECT ON THE COURSE OF COVID-19 IN ESTONIAN CHILDREN
Status: Completed | Type: Observational
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Irja Lutsar, Professor of Medical Microbiology, University of Tartu
Other Study IDs: 268/T-15
Record Dates: First submitted 2025-01-17; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: COVID - 19; Diabetes Mellitus; Post-COVID Conditions; MIS-C Associated With COVID-19
MeSH Terms: conditions — COVID-19; Diabetes Mellitus; Post-Acute COVID-19 Syndrome; pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COVID-19 children and adolescents: All the Estonian children aged <18 years with SARS-CoV-2 positivity or COVID-19 diagnosis (ICD-10 codes U07.1, U07.2)

SUMMARY:
The study focuses on Estonian children under 18 who had COVID-19 from 27.02.2020 to 01.03.2023. The main aim is to find out the risk factors for severe COVID-19 in children. In order to do that the study includes their demographic data, vaccination status, and details about the severity of illness, such as hospitalization and long-term effects of COVID-19.

DETAILED DESCRIPTION:
Data is collected for all children under 18 years old in Estonia who were diagnosed with COVID-19 between 27.02.2020 and 01.03.2024 (either with the ICD-10 codes U07.1/U07.2 and/or a positive SARS-CoV-2 test. The following data is collected for each patient: age at the time of COVID-19 diagnosis, gender, place of residence, and COVID-19 vaccination status.

In order to assess the severity of the disease, the following data is collected for each case: hospitalization due to COVID-19, length of hospitalization, need for intensive care, need for mechanical ventilation, fatal outcomes, and occurrence of long-term sequelae (post-COVID-19 condition and pediatric systemic inflammatory response syndrome). Additionally, data on any comorbid chronic and acute diseases of the children in the study group is collected. The outcome measures are compared across five different SARS-CoV-2 VOC periods: original, Alpha, Delta, Omicron BA.1/BA.2 and Omicron BA.4/BA.5.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 positivity or COVID-19 diagnosis (ICD-10 codes U07.1, U07.2)
* COVID-19 diagnosis in the following time period: 27/Feb/2020 to 01/Mar/2023

Exclusion Criteria:

* age above 18 years

Ages: 0 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All the Estonian children and adolescents (under 18 yo) who received COVID-19 diagnosis or positive SARS-CoV-2 test in a 3 year period
Sampling Method: Probability Sample
Enrollment: 127277 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Hospitalization due to COVID-19 | From enrollment to the end of the observation period in Oct 2023
  Cases requiring hospital care due to COVID-19, hospitalization length, need for intensive care
Post-COVID condition | From enrollment to the end of the observation period in Oct 2023
  Receiving post COVID-19 syndrome (ICD-10 code U09) diagnosis after acute COVID-19 infection, the time from COVID-19 to long-COVID
Diabetes mellitus | From enrollment to the end of the observation period in Oct 2023
  Receiving diabetes mellitus (ICD-10 code E10) diagnosis after acute COVID-19 infection
MIS-C | From enrollment to the end of the observation period in Oct 2023
  Receiving MIS-C diagnosis (ICD-10 code U10)
Mortality | From enrollment to the end of the observation period in Oct 2023
  Cases of COVID-19 that resulted in death

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tartu, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No
The IPD collected throughout this trial will not be shared due to data protection laws.